CLINICAL TRIAL: NCT05774444
Title: Investigating the Effects of Krill Oil and Krill Protein on Post-exercise Muscle Protein Metabolism: a Randomised Controlled Trial
Brief Title: Investigating the Effects of Krill Oil and Krill Protein on Post-exercise Muscle Protein Metabolism
Acronym: KIPLING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Aker BioMarine (Unknown)
Responsible Party: Principal Investigator, Stuart Gray, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KIPLING
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hypertrophy
Keywords: Omega-3; Krill oil; Protein; Exercise
MeSH Terms: conditions — Hypertrophy; Motor Activity | interventions — krill protein extract; Plant Oils; Carbohydrates

STUDY DESIGN:
Intervention Model Description: Parallel 2x2 factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All supplements with be colour and flavour matched
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vegetable oil + Carbohydrate (Placebo Comparator): The vegetable oil will be a placebo control for the Krill oil (4g/day). The carbohydrate will be a placebo control for the Krill protein (20g)
  Interventions: Dietary Supplement: Vegetable oil; Dietary Supplement: Carbohydrate
- Vegetable oil + Krill protein (Experimental): The vegetable oil will be a placebo control for the Krill oil (4g/day). Krill protein will be our active intervention (20g)
  Interventions: Dietary Supplement: Krill protein; Dietary Supplement: Vegetable oil
- Krill oil + Carbohydrate (Experimental): The Krill oil will be the active supplement for the intervention (4g/day). The carbohydrate will be a placebo control for the Krill protein (20g)
  Interventions: Dietary Supplement: Krill oil; Dietary Supplement: Carbohydrate
- Krill oil + Krill protein (Experimental): Both the Krill oil (4g/day) and the Krill protein will be the active intervention supplements (20g)
  Interventions: Dietary Supplement: Krill oil; Dietary Supplement: Krill protein

INTERVENTIONS:
Dietary Supplement: Krill oil — Krill oil will be supplemented to see if they can gain strength and/or muscle mass following supplementation.
  Arms: Krill oil + Carbohydrate; Krill oil + Krill protein
Dietary Supplement: Krill protein — Krill protein will be given to the participant following a resistance exercise bout.
  Arms: Krill oil + Krill protein; Vegetable oil + Krill protein
Dietary Supplement: Vegetable oil — This will be the control against the Krill oil
  Arms: Vegetable oil + Carbohydrate; Vegetable oil + Krill protein
Dietary Supplement: Carbohydrate — This will be the control for the Krill protein
  Arms: Krill oil + Carbohydrate; Vegetable oil + Carbohydrate

SUMMARY:
The aim of the current study is to find out if krill oil can increase muscle building processes in response to resistance (weightlifting) type exercise. Others aim are to determine the effects of krill protein, and the interaction of krill oil and protein, on muscle building processes in response to resistance (weightlifting) type exercise.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years old or older
* Have a BMI of less than 35kg/m2
* Be participating in structured exercise for less than 2h per week

Exclusion Criteria:

* Diabetes
* Severe cardiovascular disease
* Seizure disorders,
* Uncontrolled hypertension (>150/90mmHg at baseline measurement)
* Cancer or cancer that has been in remission <5 years
* Ambulatory impairments which would limit ability to perform assessments of muscle function
* Dementia
* Taking medication known to affect muscle (e.g., steroids)
* Have an implanted electronic device (e.g., pacemaker/defibrillator/insulin pump),
* Anticoagulant therapy
* Allergies to seafood
* Regular consumption of more than 1 portion of oily fish per week.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Post-exercise muscle protein synthesis | 3-7 hours
  Muscle protein synthesis measured 3-7h after a single bout of resistance exercise

SECONDARY OUTCOMES:
Change in Muscle thickness | Change from baseline to 8 weeks
  Vastus lateralis muscle thickness measured by ultrasound
Change in grip strength | Change from baseline to 8 weeks
  Grip strength measured with a Jamar dynamometer
Change in fat mass | Change from baseline to 8 weeks
  Whole body fat mass measured by BIA
Change in lean mass | Change from baseline to 8 weeks
  Whole body lean mass measured by BIA
Change in muscle strength | Change from baseline to 8 weeks
  Knee extensor muscle strength measured isometrically
Change in Chair rise time | Change from baseline to 8 weeks
  Time taken to get up and down from a chair 5 times
Change in balance | Change from baseline to 8 weeks
  Ability to stand for 10 seconds in full tandem, semi-tandem and feet together
Change in gait speed | Change from baseline to 8 weeks
  Time taken to walk 4 metres at a normal walking pace
Basal muscle protein synthesis | 0-3 hours
  Muscle protein synthesis measured from 0-3h after an overnight fast
Change in Erythrocyte fatty acid profile | Change from baseline to 8 weeks
  Erythrocyte fatty acid profile

CONTACTS AND LOCATIONS:
Locations (1):
- Stuart Robert Gray, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No